CLINICAL TRIAL: NCT01801397
Title: A Pilot Study to Evaluate the Effect of Forsteo (Teriparatide, 1-34-rh-PTH) in Anorexia Nervosa Patients With Low Bone Mineral Density and Increased Bone Fagility (FAN-Trial)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Psy-Rheu_2011/1
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Low Bone Mass in Anorexia Nervosa Patients

ARMS (1):
- Teriparatide (Other): one arm study. All patients receive teriparatide
  Interventions: Drug: osteoanabolic therapy

INTERVENTIONS:
Drug: osteoanabolic therapy

SUMMARY:
Study Title:

A pilot study to evaluate the effect of Forsteo® (Teriparatide, 1-34 rh-PTH) in Anorexia Nervosa patients with low mineral density and increased bone fragility (FAN-Trial)

Short Title/Study ID:

FAN-Trial / Psy-Rheu_2011/1

Indication:

Low bone mineral density (Z-Score < -1.5 or T-Score < -1.5 if available) and fragility fractures or very low bone mineral density (Z-Score < -2.5 or T-Score <-2.5 if available) without fragility fractures in Anorexia Nervosa patients

Trial Design:

Open-label, single-centre pilot study with study drug treatment duration of 24 months.

Study Center:

Single-centre (University Hospital of Zürich)

Investigator(s)/Authors:

PD Dr. med Gabriella F. Milos (Principle Investigator and author), Dept of Psychiatry, Centre for Eating Disorders, University Hospital Zürich, CH-8091 Zürich Dr. med. Diana P. Frey (Co-Investigator and author), Dept. of Rheumatology, University Hospital Zürich, CH-8091 Zürich PD Dr. med. Daniel Uebelhart (author), SUVA Fribourg, CH-1701 Fribourg

Objective(s)/Outcome(s):

Primary endpoint:

•To assess the efficacy of Teriparatide (Forsteo®) in increasing the bone mineral density in the lumbar spine, total hip and femoral neck in patients with anorexia nervosa and low bone density at months 12 and 24.

Secondary endpoints:

* To assess the changes in blood biomarkers
* To assess changes in whole body composition
* To assess the incidence of new fragility fractures
* To assess changes in bone structure
* To assess the changes in EDE-Q
* Longterm safety and tolerability of Teriparatide (Forsteo®) in patients with AN

Assessments for primary endpoint:

•BMD at lumbar spine, total hip and femoral neck, measured by DXA

Assessments for secondary endpoints:

* bone resorption and bone formation markers measured in urine and serum
* whole body composition measured by DXA
* New clinical peripheral and vertebral fractures
* HRqCT of tibia and forearm
* EDE-Q Score at months 12 and 24

Safety measurements:

* Safety lab (blood and urine)
* Clinical adverse event monitoring at all visits Number of Subjects: 10

Diagnosis and Main Inclusion Criteria:

* Women, aged > 18 to < 35 years
* Having severe anorexia nervosa (AN) (DSM-IV-R) for > 12 months before screening
* Presenting with very low bone mineral density (defined as Z-Score < -2.5 or T-Score < -2.5 if available) of at least one of the assessed localizations (lumbar spine L1 - L4, total hip, femoral neck) without any previous fragility fracture
* or low bone mineral density (defined as Z-Score < -1.5 or T-Score < -1.5 if available) of at least one of the assessed localizations (lumbar spine L1 - L4, total hip, femoral neck) and at least one previous fragility fracture
* In- and out-patients of the Centre for Eating Disorders at the Clinic for Psychiatry and Psychotherapy of the University Hospital of Zurich.

Main Exclusion Criteria:

* Metabolic bone diseases other than primary osteoporosis (including hyperparathyroidism, osteomalacia, Paget's disease of bone), pre-existing hypercalcemia, severe renal impairment (GFR < 30 ml/min), prior external beam or implant radiation therapy to the skeleton, skeletal malignancies or bone metastases, any unknown elevation of serum alkaline phosphatase, severe psychiatric diseases other than AN, drug addiction, HIV positive patients, pregnancy, open epiphyses
* Incapacity to understand the aims of the study or patients not willing to collaborate.

Study Product, Dose, Route, Regimen:

Teriparatide (Forsteo®), 20µg s.c. daily for 24 months.

Duration of study:

24 months.

Reference therapy, Dose, Route, Regimen:

NA

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria: •Women, aged > 18 to < 35 years

* Having severe anorexia nervosa (AN) (DSM-IV-R) for > 12 months before screening
* Presenting with very low bone mineral density (defined as Z-Score < -2.5 or T-Score < -2.5 if available) of at least one of the assessed localizations (lumbar spine L1 - L4, total hip, femoral neck) without any previous fragility fracture
* or low bone mineral density (defined as Z-Score < -1.5 or T-Score < -1.5 if available) of at least one of the assessed localizations (lumbar spine L1 - L4, total hip, femoral neck) and at least one previous fragility fracture
* In- and out-patients of the Centre for Eating Disorders at the Clinic for Psychiatry and Psychotherapy of the University Hospital of Zurich.

Exclusion criteria: Metabolic bone diseases other than primary osteoporosis (including hyperparathyroidism, osteomalacia, Paget's disease of bone), pre-existing hypercalcemia, severe renal impairment (GFR < 30 ml/min), prior external beam or implant radiation therapy to the skeleton, skeletal malignancies or bone metastases, any unknown elevation of serum alkaline phosphatase, severe psychiatric diseases other than AN, drug addiction, HIV positive patients, pregnancy, open epiphyses

•Incapacity to understand the aims of the study or patients not willing to collaborate.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of Teriparatide (Forsteo®) in increasing the bone mineral density in the lumbar spine, total hip and femoral neck in patients with anorexia nervosa and low bone density at months 12 and 24. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Milos, MD, Principal Investigator — University Hospital Zurich, Department of Psychiatry
Locations (2):
- Switzerland (2):
  - University Hospital Zurich, Department of Psychiatry, Zurich, Canton of Zurich
  - University Hospital Zurich, Rheumatology Department, Zurich, Canton of Zurich